CLINICAL TRIAL: NCT04498650
Title: A Phase 2b Multicentre, Randomized, Double-blind, Placebo-controlled, Parallel Group Dose Finding, Safety, Tolerability and Efficacy Study of PQ912 in Subjects With MCI and Mild Dementia Due to Alzheimer's Disease.
Brief Title: A Study to Evaluate Safety and Tolerability of Different Doses and Efficacy of PQ912 in Subjects With MCI and Mild AD
Acronym: VIVIAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vivoryon Therapeutics N.V. (Industry)
Collaborators: Nordic Bioscience A/S (Industry); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBD-01180; 2019-003532-23 (EudraCT Number)
Record Dates: First submitted 2020-07-21; First posted 2020-08-04 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Early Alzheimers Disease; Mild Cognitive Impairment Due to AD
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 300 mg (Experimental): Dose in weeks 1 and 2: 50 mg once daily (evening) Dose in weeks 3 and 4: 50 mg BID Dose in weeks 5-8: 150 mg BID Dose in weeks 9-24: 300 mg BID
  Interventions: Drug: PQ912
- 600 mg (Experimental): Dose in weeks 1 and 2: 50 mg once daily (evening) Dose in weeks 3 and 4: 50 mg BID Dose in weeks 5-8: 150 mg BID Dose in weeks 9-12: 300 mg BID Dose in weeks 12-24: 600 mg BID
  Interventions: Drug: PQ912

INTERVENTIONS:
Drug: PQ912 — PQ912 50 mg tablets and 150 mg tablets
  Other Names: varoglutamstat
  Arms: 300 mg; 600 mg
Drug: Placebo — Placebo tablets to mimic PQ912 50 mg and 150 mg tablets
  Arms: Placebo

SUMMARY:
This is a phase 2B multicenter, randomized, double-blind, placebo-controlled, parallel group dose finding study to evaluate the safety, tolerability and efficacy of PQ912, an inhibitor of the glutaminyl cyclase enzyme, in 250 subjects with mild cognitive impairment and mild dementia due to Alzheimer 's Disease.

DETAILED DESCRIPTION:
In the parallel group dose finding part of the study the first 90 subjects will be randomized 1:1:1 between PQ912 300 mg BID, 600 mg BID, and placebo. When the 90th patient has completed the week 24 treatment visit, the DSMB will decide on the dose of PQ912 to be continued. The decision is based on safety findings only, no efficacy data will be considered. After the DSMB has reached a decision on the dose to be continued, all subjects randomized to receive PQ912 will be reallocated to this dose (1:1). The duration of Subjects participation in the study is either 48, 60, 72, 84 or 96 weeks of treatment (depending on time of randomization). Subjects recruited early into the study will be kept on treatment for 96 weeks or until the regular, scheduled study visit which is closest to the scheduled week 48 visit of the last subject recruited in the study, whichever comes first.

ELIGIBILITY:
Main Inclusion Criteria:

* Positive CSF AD biomarker signature according to the AA-NIA criteria
* Clinical syndrome of MCI or mild dementia according to the AA-NIA Research Framework
* A cognitive impairment in the WAIS IV Coding Test of at least 0.5 standard deviation below the normative data
* Adequate visual and auditory abilities to perform the cognitive and functional assessments in the opinion of the investigator
* Meeting the completion and performance criteria for the CogState NTB
* Outpatient with study partner capable of accompanying the subject on all applicable clinic visits

Main Exclusion Criteria:

* Significant neurological or psychiatric disorders, other than AD, that may affect cognition.
* Atypical clinical presentations of MCI due to AD or mild dementia due to AD, such as the visual variant of AD (including posterior cortical atrophy), frontal variant or the language variant (including logopenic aphasia).
* Moderate and severe dementia with a Mini-Mental State Examination score (MMSE) below 20.
* Current presence of a clinically important major psychiatric disorder (e.g. major depressive disorder) as defined by DSM-5 criteria, or symptom(s) (e.g. hallucinations) that could affect the subject's ability to complete the study.
* History of clinically evident stroke.
* History of seizures within the last two years prior to the screening visit.
* Myocardial infarction within the last six months prior to screening.
* History of uncontrolled hypertension (in the opinion of the investigator) within six months prior to screening.
* Contraindication to lumbar puncture and MRI

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Primary safety: The proportion of participants who experience any Adverse Event (AE), Serious Adverse Event (SAE), Adverse Event of Interest (AE-I) | 48 weeks
  The safety analysis will include the number of subjects with, and the number of any AE, any SAE (both overall and related), AEs leading to discontinuation of treatment, AEs leading to temporary treatment interruption, treatment compliance, the number of subjects with AEs of interest as defined above, the severity, duration and outcome of AEs
Primary efficacy: within-participant linear change with time of the combinded z-score for cognition compared between active arm and placebo. | 48 weeks and EoT (96 weeks at maximum)
  The within-participant change over time in cognition measured by the combined z-score of the Detection test, Identification test and the 'One Back' test (attention and working memory domains) of the Neurological Test Battery

SECONDARY OUTCOMES:
Secondary efficacy: The within-participant linear change from baseline to week 48 in quantitative EEG (global relative theta wave power), compared between active and placebo. | 48 weeks at minimum or until EoT (96 weeks at maximum)
  Using a quantitative EEG the within-participant change from baseline to week 48 of the global relative theta wave power (4-8 Hz) will serve as a primary efficacy outcome.
Secondary efficacy: The within-participant linear change with time in overall cognition as measured by the CogState Brief Battery (CBB) Z-score compared between active arm and placebo | 48 weeks and EoT (96 weeks at maximum)
  he within-participant linear change with time in overall cognition as measured by the CBB (CogState Detection, Identification, One Card Learning and One Back test) -Z-score

OTHER OUTCOMES:
Exploratory efficacy - The within-participants change from baseline in a set of representative functional network topology EEG measures compared between active arms and placebo. | 48 weeks
  Evaluation of brain functional network activity and connectivity will be performed using quantitative EEG measurements, as described by (Briels et al. 2020; Poil et al. 2013; Scheltens et al. 2018) Global relative power in the delta (0.5 - 4 Hz), alpha (8 -13 Hz) and beta (13 - 30Hz) frequency bands
  * Global posterior dominant peak frequency
  * Amplitude Envelope Correlation (AEC) in the 4- 13 Hz band Functional network topology measures such as centrality, modularity, minimum spanning tree.

CONTACTS AND LOCATIONS:
Overall Officials: Everard Vijverberg, Dr, Study Chair — VUmc Alzheimer Centre
Locations (21):
- Denmark (3):
  - Sanos Clinics, Ganderup
  - Sanos Clinics, Herlev
  - Sanos Clinics, Vejle
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Schleswig-Holstein (UKSH), Klinik für Neurologie, Kiel
  - Universitätsklinikum Magdeburg / Institut für Kognitive Neurologie und Demenzforschung, Magdeburg
  - Institut für Studien zur Psychischen Gesundheit (ISPG), Mannheim
  - Klinikum rechts der Isar der TU München / Klinik für Psychiatrie und Psychotherapie, München
  - Universitätsklinikum Münster / Klinik für Allgemeine Neurologie, Münster
  - Klinik für Neurologie Universitätsklinikum Ulm, Ulm
- Netherlands (3):
  - Brain Research Center, 's-Hertogenbosch
  - Brain Research Center, Amsterdam
  - Brain Research Center Zwolle, Zwolle
- Poland (4):
  - Podlaskie Centrum, Bialystok
  - SOMED CR, Lodz
  - Klinika Psychiatrii Wieku Podeszłego i Zaburzeń Psychotycznych Uniwersytetu Medycznego w Łodzi, Lodz
  - SOMED CR, Warsaw
- Spain (4):
  - Neurology (Memory Unit) - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Fundació ACE, Barcelona
  - Cae Oroitu, Getxo
  - Unidad de Neurociencias. Hospital Victoria Eugenia, Seville

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Vijverberg EGB, Axelsen TM, Bihlet AR, Henriksen K, Weber F, Fuchs K, Harrison JE, Kuhn-Wache K, Alexandersen P, Prins ND, Scheltens P. Rationale and study design of a randomized, placebo-controlled, double-blind phase 2b trial to evaluate efficacy, safety, and tolerability of an oral glutaminyl cyclase inhibitor varoglutamstat (PQ912) in study participants with MCI and mild AD-VIVIAD. Alzheimers Res Ther. 2021 Aug 23;13(1):142. doi: 10.1186/s13195-021-00882-9. PMID 34425883